CLINICAL TRIAL: NCT05993247
Title: Efficacy of Probiotics for Non-steroidal Anti-inflammatory Drug-induced Enteropathy in Arthritis Patients: A Double-blinded Pilot Randomized Controlled Trial
Brief Title: Efficacy of Probiotics for NSAID-induced Enteropathy in Arthritis Patients
Acronym: NSAID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jae Myung Park (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor-Investigator, Jae Myung Park, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KC23MISI0269
Record Dates: First submitted 2023-07-20; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Probiotics group vs. Placebo group
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics arm (Active Comparator): Probiotics combination capsule (Bacillus Subtilis 150 mg /Clostridium Burtyricum Toa 150 mg /Saccharomyces Boulardii 113 mg) per oral, three times a day, for 8 weeks
  Interventions: Combination Product: Probiotics capsule
- Placebo arm (Placebo Comparator): Placebo capsule in the same form as probiotics, per oral, three times a day, for 8 weeks
  Interventions: Combination Product: Placebo capsule

INTERVENTIONS:
Combination Product: Probiotics capsule — Subjects will take a probiotics combination capsule (Bacillus Subtilis 150 mg /Clostridium Burtyricum Toa 150 mg /Saccharomyces Boulardii 113 mg) three times a day for 8 weeks in combination with NSAIDs
  Arms: Probiotics arm
Combination Product: Placebo capsule — Subjects will take a placebo capsule identical in shape and size to probiotics capsule three times a day for 8 weeks in combination with NSAIDs
  Arms: Placebo arm

SUMMARY:
This study aimed to investigate the efficacy of probiotics as a preventive agent for NSAID-induced enteropathy. Arthritis patients are randomly divided into probiotic and placebo groups, and the drug is administered for eight weeks. Before and after drug administration, the patient's symptoms/degree of small bowel injuries on capsule endoscopy/microbiome composition and diversity were investigated.

DETAILED DESCRIPTION:
Background:

Due to aging, there are many long-term users of NSAIDs, increasing enteropathy. The prophylactic effect of misoprostol, which is currently used, has not been proven, and misoprostol's long-term compliance and safety remain questionable. Rebamipide shows insignificant effects in both treatment and prophylaxis.

Probiotics have been reported to affect enteropathy in animal and human studies. However, there needs to be more verification studies, and there needs to be confirmatory studies on the importance of the microbiome in the small bowel. However, it is expected that there will be fewer complications and less patient resistance, resulting in higher drug compliance.

Purpose: To identify the efficacy of probiotics on NSAID-induced enteropathy in arthritis patients by capsule endoscopy and questionnaire, and to analysis the composition and diversity of the microbiome

Design: Double-blinded randomized controlled, pilot study

Participant: Patients diagnosed with osteoarthritis and starting NSAIDs

Methods: Randomly administering Probiotics or Placebo for eight weeks and comparing "before and after administration" in arthritis patients

1. Survey of patient symptoms for enteropathy
2. Recovery of small bowel mucosal injuries in capsule endoscopy
3. Analysis of the composition and diversity of the microbiome
4. Adverse events

Outcome

* Primary outcome: To assess whether probiotics can reduce small bowel injuries caused by NSAIDs
* Secondary outcome:

  1. To investigate whether probiotics can reduce gastrointestinal symptoms caused by NSAIDs
  2. To identify the improvement of arthritis symptoms
  3. To examine whether the distribution of the microbiome can be converted into beneficial bacteria by administering probiotics

ELIGIBILITY:
Inclusion Criteria:

* Patients with axial SpA who meet the 2009 ASAS criteria or osteoarthritis diagnosed by hand or foot x-rays

Exclusion Criteria:

* History of taking NSAIDs or antibiotics within the last month
* Those who have been taking probiotics, steroids, or immunosuppressants for a long time
* Abdominal surgical history (exception: appendectomy, cholecystectomy)
* History of gastrointestinal malignant disease
* Abnormal findings requiring drug treatment or surgery in upper gastrointestinal endoscopy (e.g., digestive cancer, acute peptic ulcer, etc.)
* Hemorrhagic disease
* Anemia with hemoglobin less than 10 g/dL
* Past NSAIDs drug side effects (allergy)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the small bowel injuries on capsule endoscopy | From enrollment to the end of treatment at 8 weeks
  Changes in the number of ulcers/erosions in the small bowel mucosa on capsule endoscopy before and after taking the NSAIDs and Probiotics/Placebo

SECONDARY OUTCOMES:
Change from Baseline in Gastrointestinal Symptom Rating Scale (GSRS) Questionnaire Scores | From enrollment to the end of treatment at 8 weeks
  Change from Baseline in Gastrointestinal Symptom Rating Scale Questionnaire Scores at 8 Weeks
  * Symptoms: Pain or discomfort in upper abdomen, Heartburn, Acid reflux, Hunger pangs, Nausea, Rumbling, Bloating, Passing gas, Constipation, Diarrhea, Loose stool, Hard stool, Urgent bowel movement, Sensation of not completely emptying bowel
  * Scoring: Each of the 15 items is scored from 0 to 6 points, with the highest score being 45 points and the lowest being 0 points. A score of 0 means no gastrointestinal symptoms, and a higher score indicates a more frequent occurrence of the corresponding symptoms.
Change From Baseline in Symptom Scores on the Western Ontario and McMaster Universities (WOMAC) Arthritis Index | From enrollment to the end of treatment at 8 weeks
  * WOMAC index: Descending stairs, Ascending stairs, Rising from sitting, Standing, Bending to floor, Walking on flat surface, Getting in/out of car, Going shopping, Putting on socks, Lying in bed, Talking off socks, Rising from bed, Getting in/out of bath, Sitting, Getting on/off toilet, Heavy domestic duties, Light domestic duties
  * Each of the 24 items is scored from 0 to 4 points, with the highest score being 96 points and the lowest being 0 points. A score of 0 means no symptoms and a higher score indicates more severe symptoms of the corresponding symptoms.
Change From Baseline in Symptom Scores on the Knee Injury and Osteoarthritis Outcome Scores (KOOS) Questionnaire at 8 Weeks | From enrollment to the end of treatment at 8 weeks
  * Assessment of KOOS: Daily living, Sports and recreational activities, Pain, Quality of life, Symptoms and stiffness
  * Each of the 42 items is scored from 0 to 4 points, with the highest score being 168 points and the lowest being 0 points. A score of 0 means no symptoms, and a higher score indicates more severe and frequent symptoms of the corresponding symptoms.
Changes in the gut microbiome through Next Generation Sequencing | From enrollment to the end of treatment at 8 weeks
  * Changes in composition and diversity of gut microbiota through stool samples
  * Changes in microbial genome composition

CONTACTS AND LOCATIONS:
Overall Officials: Jae Myung Park, MD, Study Chair — The Catholic University of Korea